CLINICAL TRIAL: NCT01895296
Title: Exploratory Randomized, Placebo-controlled Study to Assess Safety and Efficacy of sc Pasireotide in Patients With Dumping Syndrome
Brief Title: Study to Assess Safety and Efficacy of sc Pasireotide in Patients With Dumping Syndrome
Acronym: CSOM230BBE01T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Professor of Medicine, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSOM230BBE01T; 2008-000700-84 (EudraCT Number)
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Dumping Syndrome
Keywords: dumping syndrome; OGTT; hypoglycemia
MeSH Terms: conditions — Dumping Syndrome; Hypoglycemia | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pasireotide (Experimental): pasireotide 300 microgram s.c. t.i.d.
  Interventions: Drug: Pasireotide
- Placebo (Placebo Comparator): saline s.c. t.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pasireotide — somatostatin analogue pasireotide
  Other Names: SOM230
  Arms: Pasireotide
Drug: Placebo — placebo s.c.
  Arms: Placebo

SUMMARY:
Dumping Syndrome consists of (1) a too rapid gastric emptying, (2) an inappropriate release of GI hormones (as a reaction to the hyperosmolar contents in the duodenum) and (3) an hyperinsulinemic response to a too rapid absorption of glucose. Because it is not well known which somatostatin receptor(s) (sst1-5) influence(s) Dumping Syndrome most, the goal of this trial is to evaluate :

* the effect of pasireotide (sst1, 2, 3, 5 agonist) on the control of gastric emptying.
* the effect of pasireotide (sst1, 2, 3, 5 agonist) on the release of GI hormones (during OGTT).
* the effect of pasireotide (sst1, 2, 3, 5 agonist) on the hyperinsulimic response (during OGTT).
* the efficacy of pasireotide (sst1, 2, 3, 5 agonist) for control of objective parameters of Dumping Syndrome (hematocrit (Hct), pulse rate and occurrence of hypoglycemia after an Oral Glucose Tolerance Test (OGTT) with 75g of glucose)
* the efficacy of pasireotide (sst1, 2, 3, 5 agonist) for control of overall symptoms as measured by the combined Dumping Syndrome score
* the efficacy of pasireotide (sst1, 2, 3, 5 agonist) for control of symptoms as measured by (a) early and (b) late phase dumping symptom score separately
* the efficacy of pasireotide (sst1, 2, 3, 5 agonist) for control of quality of life (QoL SF-36)

DETAILED DESCRIPTION:
This will be a single centre, randomized, double-blind, controlled cross-over study during 35 days.

After a 4 weeks screening period, patients who fulfill the entrance criteria will be randomly assigned on a 1:1 basis to either the pasireotide treatment arm or to the placebo treatment arm. They will be treated with pasireotide sc or placebo sc for 2 weeks. After 2 weeks, patients will be switched to the other treatment arm after a 7 days wash out period. This phase is double-blind: both the patient and investigator will be blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 80 years.
* Patients with diagnosis of Dumping Syndrome:
* Having symptoms of Dumping Syndrome (sum of combined Dumping Syndrome score ≥10) AND

  * either (a) having had a documented episode of postprandial hypoglycemia in the medical history
  * or either (b) demonstrating a hypoglycemia (<60mg/dl) or hematocrite increase of > 3% or a pulse increase of 10 bpm after an oral glucose tolerance test with 75 g of glucose.
* Patients for whom written informed consent to participate in the study has been obtained. Patients will need to provide their informed consent prior to starting any medication washout period

Exclusion Criteria:

* Patients who have undergone major surgery/surgical therapy for any cause within 1 month
* Patients with symptomatic cholecystolithiasis in the medical history unless a cholecystectomy is performed (ultrasound abdomen maximum 6 months old).
* Patients who have failed treatment with somatostatin analogues in the past (specifically patients who have been treated with octreotide s.c. for more than 2 days or with a long acting somatostatin analogue for more than 8 weeks).
* Patients who have been treated with somatostatin analogues during the last 12 weeks before inclusion.
* Patients who have a known hypersensitivity to somatostatin analogues.
* Patients with the diagnosis of Diabetes Mellitus
* Patients with important co-morbidity (cardiac, pulmonary, renal , hepatic diseases)
* Patients with abnormal coagulation (PT and PTT elevated by 30% above normal limits)
* Patients receiving anticoagulants that affect PT or PTT
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control. Female patients must use barrier contraception in addition to condoms. If oral contraception is used, the patient must have been practicing this method for at least three months prior to the enrollment and must agree to continue the oral contraceptive throughout the course of the study, and for three months after the study has ended. Male patients who are sexually active are required to use condoms during the study and for 3 months afterwards.
* History of immunocompromise, including a positive HIV test result (ELISA and Western blot). A HIV test will not be required; however, previous medical history will be reviewed
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Patients with additional active malignant disease within the last five years (with the exception of basal cell carcinoma or carcinoma in situ of the cervix)
* Patients with the presence of active or suspected acute or chronic uncontrolled infection
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: symptoms related to Dumping Syndrome Severity Score | 2 weeks
  The dumping score is the sum of the early and late dumping symptoms. Early dumping starts immediately after a meal, within 1 hour (< 1 hour). Late dumping starts later than 1 hour after a meal (≥ 1 hour). In case a symptom starts immediately after a meal and lasts longer than 1 hour, the score for early AND late dumping should be ticked.
  Dumping Score None Mild Moderate Severe Early Dumping 0 1 2 3 Sweating 0 1 2 3 Flushes 0 1 2 3 Dizziness 0 1 2 3 Palpitations 0 1 2 3 Abdominal pain 0 1 2 3 Diarrhea 0 1 2 3 Bloating 0 1 2 3 Nausea 0 1 2 3
  None Mild Moderate Severe Late Dumping 0 1 2 3 Sweating 0 1 2 3 Palpitations 0 1 2 3 Hunger 0 1 2 3 Drowsiness to unconsciousness 0 1 2 3 Trembling 0 1 2 3 Irritability 0 1 2 3

SECONDARY OUTCOMES:
Effect on hypoglycemia | 2 weeks
  • The secondary efficacy variables include the proportion of patients with reduced hypoglycemic events

OTHER OUTCOMES:
Control of Hct rise | 2 weeks
  Proportion of patients with hematocrit rise during OGTT
Control of pulse rate rise | 2 weeks
  Proportion of patients with pulse rate rise during OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, M.D., Ph.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium